CLINICAL TRIAL: NCT01172340
Title: Behavioral/Support Intervention for Diet and Exercise Among Underserved Women
Brief Title: Diet and Exercise for Underserved Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Responsible Party: Principal Investigator, Patricia Sharpe, Research Professor and Co-Investigator, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00003053
Record Dates: First submitted 2010-07-28; First posted 2010-07-29 (Estimated); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Obesity
Keywords: behavioral; diet; exercise
MeSH Terms: conditions — Obesity; Behavior; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Behavioral and support intervention (Experimental): one individual counseling session with diet and exercise recommendations plus 16 weeks of group sessions, plus 8 weeks of phone followup
  Interventions: Behavioral: Behavioral and support intervention
- wait-listed control group (Placebo Comparator): Controls receive individual counseling session and recommendations, mailed health information, and after post-test measures are offered an abbreviated group-based intervention
  Interventions: Behavioral: Wait-listed control group

INTERVENTIONS:
Behavioral: Behavioral and support intervention — Individual counseling session with diet and exercise recommendations, 16 weekly group sessions, 8 weeks of followup phone support
  Arms: Behavioral and support intervention
Behavioral: Wait-listed control group — Controls receive the same individual counseling session as intervention group; receive mailed health information; are offered group sessions after last post-measure
  Arms: wait-listed control group

SUMMARY:
The purpose is to determine if a culturally tailored diet and exercise intervention of 16 weekly sessions with 8 weeks of followup phone support is effective in reducing waist circumference, weight, and related diet and exercise behaviors among women from underserved communities.

DETAILED DESCRIPTION:
Overweight and obesity disproportionately impact economically disadvantaged and minority women. Overweight and obese women ages 25 to 50 are recruited from Census tracts with 25% or more residents living below poverty-level income. A skills-based intervention was designed with input from women in these communities gathered via focus groups and from a community advisory board. The intervention activities and strategies take into consideration the social and economic challenges of women with limited income, competing demands on their time and cultural beliefs about food preferences and body image.

ELIGIBILITY:
Inclusion Criteria:

* 25-50 years of age
* live in Census tracts with 25% or more below poverty in Columbia, SC
* waist circumference >88 cm

Exclusion Criteria:

* insulin-dependent
* pregnant
* moderate exercise contraindicated
* not in control of food choices [institutional setting or restricted diet]
* uncontrolled hypertension
* weight >430 pounds

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2007-08; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
body weight | one year
  body weight in pounds is measured at baseline,16-weeks post-intervention, 24 weeks post-intervention, and at one year.
waist circumference | one year
  waist circumference in centimeters is measured at baseline,16-weeks post-intervention, 24 weeks post-intervention, and at one year.

SECONDARY OUTCOMES:
dietary fat intake | one year
  total dietary fat intake in grams and % of energy intake is assessed via 3-day dietary recall interviews at baseline,16-weeks post-intervention, 24 weeks post-intervention, and at one year.
saturated dietary fat intake | one year
  Saturated fat intake in grams and % of energy intake is measured via 3-day dietary recall interviews at baseline,16-weeks post-intervention, 24 weeks post-intervention, and at one year.
fruit and vegetable intake | one year
  Average daily servings of fruit and vegetables is measured via 3-day dietary recall interviews at baseline,16-weeks post-intervention, 24 weeks post-intervention, and at one year.
dietary fiber intake | one year
  Average daily intake of dietary fiber in grams is measured via 3-day dietary recall interviews at baseline,16-weeks post-intervention, 24 weeks post-intervention, and at one year.
total energy intake | one year
  Total energy intake in kcals is measured via 3-day dietary recall interviews at baseline,16-weeks post-intervention, 24 weeks post-intervention, and at one year.
physical activity level | one year
  Time spent in light, moderate and vigorous physical activity is estimated from 7 days of accelerometer wear at baseline,16-weeks post-intervention, 24 weeks post-intervention, and at one year.
social support | one year
  Social support for healthy eating and exercise is measure via interview at baseline,16-weeks post-intervention, 24 weeks post-intervention, and at one year.
healthy eating behaviors | one year
  Healthy eating behaviors are measured with a validated scaled via interviews at baseline,16-weeks post-intervention, 24 weeks post-intervention, and at one year.
exercise self-efficacy | one year
  Exercise self-efficacy is measured via a validated scale by interview at baseline,16-weeks post-intervention, 24 weeks post-intervention, and at one year.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia A Sharpe, PhD, MPH, Principal Investigator — University of South Carolina
Locations (1):
- Prevention Research Center, University of South Carolina, Columbia, South Carolina, United States